CLINICAL TRIAL: NCT00362440
Title: A Combination of Insulin Sensitizer and Leptin as Treatment for the HAART -Induced Metabolic Syndrome: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Combination of Insulin Sensitizer and Leptin as Treatment for the HAART -Induced Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005P000159
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: HIV Lipodystrophy
Keywords: HIV lipodystrophy; Leptin; Fat wasting; Pioglitazone; Insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Leptin; Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leptin (Experimental): Leptin replacement therapy
  Interventions: Drug: Leptin; Drug: Pioglitazone or metformin
- Pioglitazone or metformin (Placebo Comparator): Diabetes treatment therapy
  Interventions: Drug: Pioglitazone or metformin; Drug: Placebo

INTERVENTIONS:
Drug: Leptin
  Arms: Leptin
Drug: Pioglitazone or metformin
Drug: Placebo
  Arms: Pioglitazone or metformin

SUMMARY:
The purpose of this study is to determine whether patients with HIV lipodystrophy (fat wasting) benefit from taking the combination of two drugs, one insulin sensitizer (either metformin or pioglitazone, both diabetes drugs) and leptin (a natural hormone produced by your fat cells). Our hope is that they will improve sugar and fat metabolism and positively affect the body fat changes you have noticed while taking HAART.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) induces profound and sustained suppression of human immunodeficiency virus (HIV) replication, and is thus very effective in reducing disease-associated morbidity and mortality in this patient population. However, HAART also results in the development of a lipodystrophic syndrome which is characterized by fat accumulation, fat wasting, or a combination of both, and similar to congenital forms of lipodystrophy, is associated with components of the metabolic syndrome, including insulin resistance (IR), fasting hypertriglyceridemia, and hypercholesterolemia.

Our study is a "proof of concept" study on the treatment of the HAART-induced metabolic syndrome, which builds upon and represents a direct extension of a study previously funded by the American Diabetes Association (ADA). If our clinical trial proves that a combination treatment of leptin and an insulin sensitizer has additive or synergistic effects in reversing the metabolic abnormalities of HIV positive patients with lipoatrophy, it could lead to the design of larger multi-center, randomized, placebo-controlled trial(s) aiming at establishing safety and efficacy of this treatment for the HAART-induced metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age18 years and above and ability and willingness to give written informed consent
* Documented HIV-1 infection
* At least 6 months of stable cumulative antiretroviral therapy with any available or investigational anti- retroviral medication (protease inhibitor, nucleoside reverse transcriptase inhibitor, non-nucleoside reverse transcriptase inhibitor, nucleotide reverse transcriptase inhibitor)
* Lipoatrophy developed after initiating HAART treatment (see criteria below). Leptin levels should be less than 4 ng/ml.
* Insulin resistance, impaired fasting glucose, impaired glucose tolerance or type 2 diabetes developed after starting the antiretroviral medications. These categories are defined, respectively, as fasting insulin level above 15 µIU/ml; fasting serum glucose value above 100 mg/dl; 2-hour serum glucose level during a 75 gram oral glucose tolerance test (OGTT) between 140 and 200 mg/dl; and fasting glucose above 126 mg/dl or random glucose level above 200 mg/dl with presence of the classic symptoms of diabetes, such as polyuria, polydipsia, ketonuria, and rapid weight loss
* Hypertriglyceridemia and/or hypercholesterolemia developed after starting the antiretroviral therapy. These categories are defined as fasting triglycerides greater than 150 mg/dl and LDL cholesterol greater than 130 mg/dl, respectively
* Female subjects must have a negative urine pregnancy test before enrollment and must agree to use a barrier contraception i.e. condoms, diaphragm or IUD, with or without a hormonal-based method for the duration of the study. Women who are pregnant or become pregnant during the study and who do not accept some form of contraception will be excluded from the study.
* Patients should have history of peripheral fat wasting of the face (e.g. sunken cheeks), limbs (including prominent veins), and/or buttocks, which developed after the initiation of HAART therapy
* Patients should have physical exam findings of a) facial atrophy - sunken cheeks, sunken temporal regions, and/or prominent temporal veins and b) wasting of fat in periphery, limbs and/or buttocks (including prominent veins)
* Patients should have anthropometric measurements suggestive of decreased subcutaneous fat content: Decreased triceps skinfold thickness (< 4 mm in men and < 8 mm in women) or Decreased upper arm circumference (< 27.1 cm in men and < 23.3 cm in women) or Decreased subscapular skinfold thickness (< 7 mm in men and < 7 mm in women) or dual energy X-ray absorptiometry (DEXA) scanning suggestive of fat depletion: total body fat < 14% in men and < 22% in women.

Exclusion Criteria:

* History of impaired glucose metabolism or hyperlipidemia prior to antiretroviral use
* Triglyceride levels higher than 1500 mg/dl after the 1 month run-in phase or anytime during the study
* Abnormal hepatic function: liver function tests higher than twice the upper normal range
* Abnormal renal function: creatinine higher than 1.3 mg/dl
* Any condition/illness that may affect study outcomes such as pregnancy, active infection except HIV, clinically significant malabsorption/malnutrition, malignancy
* Any active hormonal disease and/or hormonal treatment that may affect the outcomes of interest such as clinically overt hypo/hyperthyroidism, hypogonadism, hypercortisolism, or treatment with steroids or growth hormone (exception: patients taking testosterone can be included in the trial if they agree to continue the same dosage for the duration of the trial)
* Present alcoholism or drug abuse. These conditions will be screened for by a detailed history and systems review and baseline laboratory analysis with chemistries, CBC, and hormone levels, and EKG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-08; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lee JH, Chan JL, Sourlas E, Raptopoulos V, Mantzoros CS. Recombinant methionyl human leptin therapy in replacement doses improves insulin resistance and metabolic profile in patients with lipoatrophy and metabolic syndrome induced by the highly active antiretroviral therapy. J Clin Endocrinol Metab. 2006 Jul;91(7):2605-11. doi: 10.1210/jc.2005-1545. Epub 2006 Apr 24. PMID 16636130

RESULTS

PARTICIPANT FLOW:
Groups:
- Leptin: Leptin replacement therapy
  Leptin+pioglitazone
- Pioglitazone or Metformin: Diabetes treatment therapy
  Pioglitazone+placebo
Period: Overall Study
Arm/Group | Leptin | Pioglitazone or Metformin
Started | 5 | 4
Completed | 3 | 3
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leptin | Pioglitazone or Metformin | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [43 to 57] | 50 [43 to 57] | 50 [43 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance (HOMA Index)
Time Frame: At the end of each 3 month intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Leptin | Pioglitazone or Metformin
Number analyzed (Participants) | 5 | 4
units on a scale | 1.6 (0.5) | 1.8 (0.8)

2. Secondary Outcome: Cholesterol Levels
Time Frame: At the end of each 3 month intervention
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Leptin | Pioglitazone or Metformin
Number analyzed (Participants) | 5 | 4
mg/dl | 190 (13) | 183 (17)

3. Secondary Outcome: Body Composition (Fat Mass)
Time Frame: At the end of each 3 month intervention
Measure: Mean (Standard Error); unit: kg
Arm/Group | Leptin | Pioglitazone or Metformin
Number analyzed (Participants) | 5 | 4
kg | 16.7 (1.7) | 13.1 (0.8)

ADVERSE EVENTS:
Arm/Group | Leptin | Pioglitazone or Metformin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leptin (N=5) | Pioglitazone or Metformin (N=4)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No